CLINICAL TRIAL: NCT02492607
Title: Management of Low Risk Ductal Carcinoma in Situ (Low-risk DCIS): a Non-randomized, Multicenter, Non-inferiority Trial; Standard Therapy Approach Versus Active Surveillance
Brief Title: Management of Low-risk (Grade I and II) DCIS
Acronym: LORD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Borstkanker Onderzoek Groep (Network); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M18LORD; 2014-04 (Other: BOOG); EORTC-1401 (Other: EORTC)
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2025-01

CONDITIONS: DCIS
Keywords: Women; DCIS grade I and II; Active surveillance; Standard treatment
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Mammography; Observation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Standard treatment according to local policy. This can be either wide local excision only, wide local excision and radiotherapy, or mastectomy. Hormonal therapy is also allowed.
  Follow-up:by annual digital mammography for a period of 5 years and a digital mammography at 7 and 10 years.
  Interventions: Other: Standard treatment; Radiation: radiotherapy
- Active surveillance (Experimental): Active surveillance : monitoring by annual digital mammography for a period of 5 years and a digital mammography at 7 and 10 years.
  Interventions: Device: digital mammography

INTERVENTIONS:
Other: Standard treatment — wide local excision only or wide local excision and radiotherapy or mastectomy.
  +/- hormonal therapy
  Arms: Standard treatment
Device: digital mammography — annual mammography
  Other Names: Active surveillance
  Arms: Active surveillance
Radiation: radiotherapy — according local policy
  Arms: Standard treatment

SUMMARY:
A substantial number of DCIS lesions will never form a health hazard, particularly if it concerns slow-growing low-risk DCIS (grade I and II). This implies that many women might be unnecessarily going through intensive treatment resulting in a decrease in quality of life and an increase in health care costs, without any survival benefit.

The LORD (LOw Risk DCIS) study is a non-randomized, international, multicenter, phase III non-inferiority trial, and aims to determine whether screen-detected low-risk DCIS can safely be managed by an active surveillance strategy or that the conventional treatment, being either WLE alone, WLE + RT, or mastectomy, and possibly HT, should remain the standard of care.

DETAILED DESCRIPTION:
Background of the study:

The introduction of population-based breast cancer screening and implementation of digital mammography have led to an increased incidence of ductal carcinoma in situ (DCIS) without a decrease in the incidence of advanced breast cancer. This suggests DCIS overdiagnosis exists. We hypothesize that asymptomatic, low-risk DCIS (grade I and II DCIS) can safely be managed by active surveillance. If progression to invasive breast cancer would still occur, this will be lowgrade and hormone receptor positive with excellent survival rates. Also, breast-conserving treatment will still be an option, if no prior radiotherapy has been applied. It also may save many low-risk DCIS patients from intensive treatment.

Objective of the study:

The primary end-point is ipsilateral invasive breast tumor-free rate at 10 years.

Secondary end-points are among others: overall survival, breast cancer-specific survival, mastectomy rate and patient reported outcomes. To determine whether low- risk DCIS can safely (measured by ipsilateral invasive breast cancer rate at 10 years) be managed by an active surveillance strategy or if the conventional treatment, being either wide local excision (WLE) only, WLE plus radiotherapy or mastectomy, possibly followed by hormonal therapy, will remain the standard of care.

Study design:

Phase III, open-label, non-inferiority, multi-center, non-randomized clinical trial. By patient's preference, women will be included into one of the following arms: active surveillance or standard treatment according to local policy, being either WLE alone, WLE plus radiotherapy or mastectomy, possibly followed by hormonal therapy. The same follow-up scheme will be applied in both study arms, i.e. annual mammography for a period of five years and an additional two mammograms at year seven and ten.

ELIGIBILITY:
Inclusion criteria

* Written informed consent according to ICH GCP, and national andlocal regulations
* Women ≥ 45 years old, any menopausal status
* Unilateral DCIS grade I or II of any size
* American Society of Anesthesiologists (ASA) score 1-2 or 3, only if able to undergo surgery and yearly mammography
* Lesions of type 'calcifications only', detected by population-based or opportunistic screening mammography
* Within twelve weeks of detection, stereotactic biopsy has to be performed from the area of the calcifications. Preferably vacuum assisted biopsies. Alternatively, at least six 12 G needle biopsies (or the equivalent of six 12 G needles) may be used. ) . Whatever needle size is applied, it is essential to confirm that the biopsies contain representative calcifications via biopsy radiography, microscopy, or both.
* Estrogen receptor ≥ 80% positive and HER2 negative: 0 or 1+ or 2+ with negative ISH), analysed centrally by pathology at NKI-AVL
* In case of an extended lesion (> 5 cm): biopsies were taken from the center and the periphery of the lesion, or from two peripheral parts of the lesion
* In case of multiple lesions with calcifications biopsies have been taken from two, but not more, groups of calcifications
* Marker placement at biopsy site (s) in the breast
* FFPE tissue blocks from the biopsy and, if applicable, from the resection specimen, are available for translational research purposes. If no FFPE tissue blocks can be submitted, 10 unstained slides of 4-5 micrometer thickness from the lesion(s) are acceptable
* Good correlation between pathological and radiological findings i.e. both findings confirm low-risk DCIS and no suspicion of high- grade DCIS or invasive breast cancer
* The interval between histologic diagnosis of low-risk DCIS on biopsy and inclusion is ≤ 12 weeks

Exclusion criteria

* Estrogen receptor negative: <80% or HER2 positive: 3+, or 2+ with positive ISH
* Presence of either mass, increased focal density or architectural distortion around the calcifications on mammography (suspicious for invasive disease)
* Presence of Paget's disease, invasive breast cancer, or pleomorphic LCIS; Lobular neoplasia, referring to atypical lobular hyperplasia (ALH) and/or classic Lobular Carcinoma In Situ according to the WHO Classification of Tumours of the Breast, is no reason to exclude, whereas pleomorphic LCIS is
* Symptomatic DCIS e.g. DCIS detected by palpation or bloody nipple discharge
* Synchronous invasive carcinoma in the contralateral breast
* Prior history of invasive breast cancer or DCIS, prior surgery because of benign breast lesion (s) is allowed
* Prior history of other malignancy (except non-melanoma skin cancer and carcinoma in situ of the cervix) unless patient is discharged from follow-up for at least five years.
* Serious disease that precludes definitive surgical treatment (e.g cardiovascular/ pulmonary/ renal disease)
* Individual with a family member with a known gene mutation associated with increased risk of breast cancer, unless study participant is a proven non-carrier of mutation
* Pregnancy or breast-feeding. Contraceptive measures during the trial are mandatory for those patients that will participate in standard treatment arm and adequate counseling should be provided by the treating physician. The duration of contraception will be specified by the treating physician according to patient and treatment characteristics, standard clinical practice and national regulations
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2034-02-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral invasive breast cancer-free rate at 10 years | 10 years from inclusion
  Ipsilateral invasive breast cancer-free rate at 10 years (both therapeutic policies

SECONDARY OUTCOMES:
Rate of invasive disease at the final pathology specimen (standard arm only) | from inclusion till time of invasive disease during 10 years at minimum
  Rate of invasive disease at the final pathology specimen (standard arm only)
Rate of grade III DCIS at the final pathology specimen (standard arm only) | from inclusion till time of invasive disease during 10 years at minimum
  Rate of grade III DCIS at the final pathology specimen (standard arm only)
Biopsy rate for ipsilateral breast during follow-up | from inclusion to the time of death, during 10 years at minimum
  Biopsy rate for ipsilateral breast during follow-up (both therapeutic policies)
Masectomy rate for ipsilateral breast | from inclusion to the time of ipsilateral breast cancer or death, during 10 years at minimum
  Masectomy rate for ipsilateral breast, baseline or subsequent ipsilateral DCIS or iBC (both therapeutic policies)
Time to ipsilateral grade III DCIS | from inclusion to the development of a new ipsilateral DCIS of grade III, up to 10 years
  Time to ipsilateral grade III DCIS, both therapeutic policies
Time to contralateral DCIS | from inclusion to the development of a new contralateral DCIS I,II,III, up to 10 years
  Time to contralateral DCIS, both therapeutic policies
Time to contralateral invasive breast cancer | from inclusion to the development of a contralateral invasive breast cancer, up to 10 years
  Time to contralateral invasive breast cancer,, both therapeutic policies
Time to failure of active surveillance strategy | from inclusion to the time patients received standard treatment to the ipsilateral breast, up to 10 years
  Time to failure of active surveillance strategy, i.e. time to crossover to standard treatment, due to any cause
Distant metastases free interval | from inclusion to the time of invasive distant metastases or death due to breast cancer, up to 10 years
  Distant metastases free interval,both therapeutic policies
Overall survival | from inclusion to the time of death, during 10 years at minimum
  Overall survival,both therapeutic policies
Health Related Quality of life | 6 times from inclusion to 10 yrs follow-up
  General QoL/global health perception, specific funcionalities, pain ( both therapeutic policies
Cost-effectiveness | 6 times from inclusion to 10 years follow-up
  Health economic evaluation (both therapeutic policies)

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Wesseling, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (60):
- Netherlands (60):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep- site Alkmaar, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Wilhelmina Ziekenhuis Assen, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Alexander Monro Ziekenhuis, Bilthoven
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente Ariensplain, Enschede
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Universitair Medisch Centrum Groningen, Groningen
  - Spaarne Gasthuis, Haarlem
  - Saxenburgh Medisch Centrum, Hardenberg
  - Ziekenhuis St. Jansdal, Harderwijk
  - Tjongerschans Ziekenhuis, Heerenveen
  - Zuyderland Medisch Centrum, Heerlen
  - Ziekenhuisgroep Twente, Hengelo
  - Ter Gooi, Hilversum
  - Spaarne ziekenhuis, Hoofddorp
  - Treant Zorggroep Bethesda, Hoogeveen
  - Dijklander, Hoorn
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Alrijne Ziekenhuis, Leiderdorp
  - Haaglanden MC Antoniushove, Leidschendam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Dijklander, Purmerend
  - Erasmus Medisch Centrum, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Franciscus Gasthuis en Vlietland, Schiedam
  - Zuyderland Ziekenhuis, Sittard
  - Antonius Ziekenhuis, Sneek
  - Zorgsaam Zeeuws-Vlaanderen, Terneuzen
  - Zorgsaam Ziekenhuis, Terneuzen
  - HagaZiekenhuis, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - St. Elisabeth Ziekenhuis, Tilburg
  - Bernhoven Ziekenhuis, Uden
  - Diakonessenhuis, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Maxima Medisch Centrum - Locatie Veldhoven, Veldhoven
  - VieCuri - Medisch Centrum voor Noord-Limburg - Locatie Venlo, Venlo
  - St Jans Gasthuis, Weert
  - Streekziekenhuis Koningin Beatrix, Winterswijk
  - Zaans Medisch Centrum, Zaandam
  - Haga ziekenhuis loc Zoetermeer, Zoetermeer
  - Gelre ziekenhuizen, Zutphen
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elshof LE, Tryfonidis K, Slaets L, van Leeuwen-Stok AE, Skinner VP, Dif N, Pijnappel RM, Bijker N, Rutgers EJ, Wesseling J. Feasibility of a prospective, randomised, open-label, international multicentre, phase III, non-inferiority trial to assess the safety of active surveillance for low risk ductal carcinoma in situ - The LORD study. Eur J Cancer. 2015 Aug;51(12):1497-510. doi: 10.1016/j.ejca.2015.05.008. Epub 2015 May 26. PMID 26025767